CLINICAL TRIAL: NCT02335047
Title: The Putative Correlation Between Impaired Hip Flexor Passivity and Common Lower Back Pain: a Pilot Study.
Brief Title: Investigation of the Putative Correlation Between Involuntary Psoas Activity During Passive Flexion of the Trunk at the Hips
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5898
Record Dates: First submitted 2014-12-15; First posted 2015-01-09 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Lower Back Pain
Keywords: reliability; clinical test; physical therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lower back pain (Other)
  Interventions: Other: Impaired passivity test

INTERVENTIONS:
Other: Impaired passivity test — Description of the test: the subject lies in the supine position on an exercise mat with his/her feet together. The subject is told to let his/her arms rest loosely by his/her side (as if they were ropes) and to keep the head aligned with the back. The examiner pulls the subject into the sitting position by pulling on the subject's wrists, with passive flexion of the trunk until the hip joint is fully flexed..

SUMMARY:
Passive flexion of the trunk (relative to the legs) may be accompanied by contraction of the psoas muscles, even when the subject has been told not to contract any muscles. The psoas contraction is involuntary and cannot be controlled by the subject. This lack of passivity might be concomitant with lower back pain: the impairment may be present when lower back pain is present and/or absent when lower back pain is absent.

The study's primary objective is thus to determine the sensitivity and/or specificity of a clinical test for impaired hip flexor passivity in cases of lower back pain during passive flexion of the trunk (from the supine position,).

The secondary objective is to show that a negative test (after administration of correcting measures) is correlated with a decrease in pain (i.e. pain intensity and the functional repercussions of pain).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30
* Social security coverage
* Ability to understand the study's objectives, procedures and risks and to provide informed, written consent
* Having been informed about the results of the prior clinical examination.

Exclusion Criteria:

* Past or concomitant infectious or cancerous diseases of the spine
* Vertebral osteosynthesis
* Acute neck or arm pain (recurrent dislocations of the glenohumeral joint, trauma in the previous 12 months, etc.)
* Lower back pain with irradiation of pain below the buttocks
* Known specific lower back pain or pain for which a differential diagnosis suggests an inflammatory, traumatic, cancerous or infectious cause
* Subjects under legal guardianship
* Known pregnancy
* Simultaneous participation in another biomedical research study of a drug or medical device.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Qualitative evaluation of impaired psoas muscle passivity during passive flexion of the trunk at the hips (while sitting). | Visit 1 (Day 0)

SECONDARY OUTCOMES:
- A visual analog scale for pain | - Visit 0 (Day 0: inclusion visit)

CONTACTS AND LOCATIONS:
Overall Officials: Mutter Catherine, MD, Principal Investigator — Les Hôpitaux universitaires de Strasbourg